CLINICAL TRIAL: NCT02110667
Title: Evaluation Of Transperineal Ultrasound For Image Guidance In The Treatment Of Prostate Cancer in Men Following Prostatectomy
Status: Completed | Type: Observational
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, H. James Wallace, MD, Medical Director, Radiation Oncology, University of Vermont Medical Center
Other Study IDs: M14-170
Record Dates: First submitted 2014-03-27; First posted 2014-04-10 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer; Post-Prostatectomy
Keywords: Prostate cancer; Prostatectomy; Ultrasound; TPUS
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prostate cancer, post-prostatectomy
  Interventions: Device: Transperineal Ultrasound

INTERVENTIONS:
Device: Transperineal Ultrasound
  Other Names: Elekta, Ltd. probe

SUMMARY:
This study is being done to find out if transperineal ultrasound (TPUS) can help define the prostate bed for radiation treatment planning and improve upon current methods of image guidance for the treatment of prostate cancer. For the patient, TPUS involves the placement of an ultrasound probe on the perineum, the skin between the scrotum and anus, while they are lying on their back in the position they will receive their treatment. Image-guidance is required for the treatment of prostate cancer because the prostate bed shifts position depending on how full the bladder and rectum are. Image-guided radiation therapy has been done at Fletcher Allen Health Care for approximately three years. Most commonly, transabdominal ultrasound images are obtained every day and compared to an ultrasound that was done on the day of treatment planning. Adjustments in radiation field position can be done on a daily basis by comparing these images. Transperineal ultrasound has never been used for image-guidance. We completed two phases of an earlier study and have developed a TPUS device and process that allow us to get clear ultrasound pictures of the prostate gland, and now we would like to explore imaging the prostate bed left after radical prostatectomy.The TPUS has three potential advantages over the transabdominal method we currently use:

1. Transabdominal ultrasound can be a challenge for some men. A full bladder helps us get clearer images, however it is difficult for some men with prostate cancer to comfortably keep a full bladder. It is also particularly difficult to get good images in larger men who have long distances from the skin surface to the prostate bed. TPUS is not dependent on a man having a full bladder and should be less dependent on the size of the man.
2. TPUS images and the planning CT images can be acquired simultaneously. This is not possible with the abdominal probe because it gets in the way of the CT machine. Simultaneous imaging eliminates the possibility of the prostate bed shifting positions during the time between imaging studies.
3. TPUS can be in place and acquire images during patient treatment (the abdominal probe gets in the way of the treatment machine) and may in the future allow us to watch the prostate bed during treatment. If we discover that we can accurately view the prostate bed in real time, TPUS may ultimately allow us to treat even smaller radiation fields and possibly decrease the risk of radiation complications.

Patients in this study will be treated for their prostate cancer with the standard image guidance technique used at Fletcher Allen Health Care: transabdominal ultrasound. In addition, one TPUS scan will be acquired at the time of the initial simulation.

To summarize, the two objectives of this study are:

1. To determine if TPUS can acquire usable, clinically pertinent IGRT images of the prostate bed.
2. To preliminarily compare TPUS images of the prostate bed to images obtained with CT and TAUS.

ELIGIBILITY:
Inclusion Criteria:

* Male, over age 18
* Clinical diagnosis of prostate cancer
* Post- prostatectomy surgery
* Undergoing external beam radiation

Exclusion Criteria:

* Unable to tolerate transperineal ultrasound

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: University of Vermont Medical Center- Radiation Oncology Patient Prostate cancer w/ prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2014-04; Primary Completion 2016-01 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The concluding outcome measure will be "number of patients with image quality equivalent to or better than CT Imaging | One measurement will be done at the time of the initial simulation. The participants will then have 8 weeks of standard external beam radiation.
  On Day 1, patients will be simulated with transabdominal ultrasound, and a treatment plan will be made employing this ultrasound as a reference point for the daily scans to be performed throughout treatment. A transperineal ultrasound will take place on Day 1 as well. The treatments will begin about 4 weeks later and take place daily for approximately 8 weeks. 3 times (each about 2 weeks apart) throughout the 8 weeks, an additional transperineal ultrasound will be performed as well. A radiation oncologist (HJW) will qualitatively describe and compare the visibility of the prostate bed, bladder, rectum, and penile bulb based on CT, TPUS and TAUS images. The prostate bed for the purposes of this study will be defined as the wall of the base of the bladder that extends from the most posterior edge of the pubic symphysis posteriorly 5 cm. We have adapted a previously used scoring system for the purposes of this study.

CONTACTS AND LOCATIONS:
Overall Officials: James Wallace, MD, Principal Investigator — Fletcher Allen Healthcare
Locations (1):
- Radiation Oncology, Fletcher Allen Healthcare, Burlington, Vermont, United States